CLINICAL TRIAL: NCT03920891
Title: Cryoballoon Pulmonary Vein Isolation vs. Radiofrequency Pulmonary Vein Isolation With Additional Right Atrial Linear Ablation for Valvular Atrial Fibrillation: Prospective Randomized Trial (CRAVA Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0141
Record Dates: First submitted 2019-04-14; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Valvular Atrial Fibrillation
Keywords: Valvular Atrial fibrillation; Radiofrequency Pulmonary vein isolation; Cryoballoon Pulmonary Vein isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon Pulmonary Vein isolation (Experimental): 1. Pulmonary vein isolation will be performed using a cryoballoon catheter.
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. A 28mm second or third cryoballoon catheter will be used.
  4. Esophageal temperature will be monitored to prevent esophageal injury.
  5. Cryoablation will be performed for 180 secs at -45°C or below on condition that the pulmonary vein is occluded with a cryoballoon.
  6. CMAP (compound motor action potential) monitoring will be done to avoid phrenic nerve damage during the freezing of the right superior pulmonary vein.
  7. The procedure and cryoablation times will be evaluated.
  8. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: Cryoballoon Pulmonary Vein isolation
- Radiofrequency Pulmonary Vein isolation (Active Comparator): 1. Pulmonary vein isolation will be performed using a radiofrequency catheter.
  2. Additional left atrium posterior wall isolation, left atrium anterior wall linear ablation, cavo-tricuspid isthmus ablation, superior vena cava-right atrial septal ablation.
  3. If any other trigger came from beyond pulmonary vein is detected after the administration of isoproterenol, additional local radiofrequency ablation will be followed.
  4. Evaluated the procedure and radiofrequency ablation time.
  5. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: Radiofrequency Pulmonary Vein isolation and Additional Right Atrial linear ablation

INTERVENTIONS:
Procedure: Cryoballoon Pulmonary Vein isolation — 1. Pulmonary vein isolation will be performed using a cryoballoon catheter.
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. A 28mm second or third cryoballoon catheter will be used.
  4. Esophageal temperature will be monitored to prevent esophageal injury.
  5. Cryoablation will be performed for 180 secs at -45°C or below on condition that the pulmonary vein is occluded with a cryoballoon.
  6. CMAP (compound motor action potential) monitoring will be done to avoid phrenic nerve damage during the freezing of the right superior pulmonary vein.
  7. The procedure and cryoablation times will be evaluated.
  8. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: Cryoballoon Pulmonary Vein isolation
Procedure: Radiofrequency Pulmonary Vein isolation and Additional Right Atrial linear ablation — 1. Pulmonary vein isolation will be performed using a radiofrequency catheter.
  2. Additional left atrium posterior wall isolation, left atrium anterior wall linear ablation, cavo-tricuspid isthmus ablation, superior vena cava-right atrial septal ablation.
  3. If any other trigger came from beyond pulmonary vein is detected after the administration of isoproterenol, additional local radiofrequency ablation will be followed.
  4. Evaluated the procedure and radiofrequency ablation time.
  5. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: Radiofrequency Pulmonary Vein isolation

SUMMARY:
Cryoballoon ablation is proven to be effective in pulmonary vein isolation in patients with paroxysmal and persistent atrial fibrillation. We previously reported that the rhythm outcome of radiofrequency (RF) catheter ablations are equivalent in patients with non-valvular atrial fibrillation and in those with surgically and hemodynamically corrected valvular atrial fibrillation. In contrast, the Cryoballoon ablation can reduce the procedure times, it cannot conduct empirical linear ablation or extra-pulmonary vein foci ablation. The aim of this study is to compare Cryoballoon pulmonary vein isolation and RF ablation including linear ablation or extra-pulmonary vein foci ablations in patients with hemodynamically corrected valvular atrial fibrillation.

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (cryoballoon PV isolation group vs. Radiofrequency Pulmonary Vein isolation and Additional Right Atrial linear ablation) (Using the Python program, a random number module is imported with the import random syntax, and the random number table for the two groups is created.)
2. Target number of subjects: 154 (77 per group)
3. Rhythm FU : 2012 ACC/AHA/ESC guidelines (Holter monitoring at the baseline, 3,6 month, and thereafter every 6 months to 24 month, then every 1 year; ECG if the patient has any symptom)
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Follow-up at 1 weeks, 3,6 months, and thereafter every 6-month after procedure.
3. Rhythm control at 3, 6 months, and thereafter every 6 months for 2 years, and every year after 2 years follow-up with Holter
4. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

C. Follow-up All the patients will be followed-up at 1 weeks, 3, 6 months, and thereafter every 6 months. If the patient shows any symptom within the clinical study period, patient will visit the outpatient clinic. ECG will be performed at every outpatient visits, and 24-hour Holter or event recording will be performed 3, 6 months, and thereafter every 6 months for 2 years, and every year after 2 years (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines). If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed in 12-lead ECG or Holter, it will be evaluated as recurrence. Recurrence within 3 months after the procedure will be classified as early recurrence, and that after 3 months will be classified as clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient with hemodynamic corrected valvular atrial fibrillation who is scheduled for ablation procedure and ≥20 and ≤80 years of age
* 2. Left atrium size < 50mm
* 3. paroxysmal atrial fibrillation that is recurrence during antiarrhythmic drug treatment or is not able to use an antiarrhythmic drug.
* 4. Patient who is indicated for anticoagulation therapy (for prevention of cerebral infarction)

Exclusion Criteria:

* 1. Patients with permanent atrial fibrillation
* 2. Atrial fibrillation associated with severe cardiac malformation or a structural heart disease that is hemodynamically affected
* 3. Patients with severe renal impairment or CT imaging difficulty using contrast media
* 4. Patients with a past history of radiofrequency ablation for atrial fibrillation or other cardiac surgery
* 5. Patients with active internal bleeding
* 6. Patients with contraindications for anticoagulation therapy(for prevention of cerebral infarction) and antiarrhythmic drugs
* 7. Patients with non-valvular atrial fibrillation
* 8. Patients with a severe comorbid disease
* 9. Expected survival < 1 year
* 10. Drug addicts or alcoholics
* 11. Patients who cannot read the consent form (illiterates, foreigners, etc.)
* 12. Other patients who are judged by the principal or sub-investigator to be ineligible for participation in this clinical study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Procedure-related cardiac complication rate | within 30 days post procedure
  including open cardiac surgery, cerebral infarction, pericardial effusion or cardiac tamponade, hematoma in the inguinal puncture site and vascular complications within 30 days post procedure
Efficacy evaluation: clinical recurrence rate | Within 1 year after 3 months of procedure
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after 3 months within 1 year; based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 3 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms

SECONDARY OUTCOMES:
Comparison of procedure time | immediate after procedure
Comparison of ablation time | immediate after procedure
Comparison of hospitalization period | immediate after procedure
Comparison of re-hospitalization rate after the procedure | immediate after procedure
Comparison of re-hospitalization rate after the procedure | 12 months after procedure
Comparison of number of electrical cardioversion after the procedure | immediate after procedure
Comparison of number of electrical cardioversion after the procedure | 12 months after procedure
Major cardiovascular event rate - death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure | immediate after procedure and 12 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea